CLINICAL TRIAL: NCT03718117
Title: CHARACTERISTICS OF ADULT PATIENTS TREATED WITH CRIZOTINIB FOR ADVANCED NON-SMALL-CELL LUNG CANCER (NSCLC) WITH ALK GENE REARRANGEMENT OR ROS1 GENE REARRANGEMENT IN GENERAL HOSPITALS.
Brief Title: Descriptive Observational Study ALK-2016-CPHG
Acronym: ALK2016CPHG
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: French College of General Hospital Pneumologists (CPHG) (Other)
Responsible Party: Sponsor
Other Study IDs: A8081060; ALK-2016-CPHG (Other: Alias Study Number)
Record Dates: First submitted 2018-03-05; First posted 2018-10-24 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-06

CONDITIONS: NSCLC; Crizotinib; ALK Gene Rearrangement or ROS1 Gene Rearrangement
Keywords: Non-Small Cell Lung Cancer (NSCLC); crizotinib; ALK gene rearrangement or ROS1 gene rearrangement
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Descriptive Observational Study.

Characteristics Of ALK-positive and ROS1-positive Adults Patients Non-Small Cell Lung Cancer (NSCLC) Treated With Crizotinib Within General Hospitals

DETAILED DESCRIPTION:
Describe the characteristics of patients treated with crizotinib Describe efficacy, safety, observance and QoL.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years
* Locally advanced or metastatic NSCLC
* Patient ALK gene rearrangement or ROS1 gene rearrangement
* Patient having initiated in the previous 3 months or patient initiating crizotinib treatment regardless of the line of treatment
* Patient followed up by a physician in a hospital pulmonary medicine department
* Subject of reproductive age, using an effective method of contraception
* Patient informed verbally and in writing on the study and having consented to his/her personal data being collected within the scope of the study.

Non-inclusion criteria

* Patient included within the scope of an interventional therapeutic trial
* Patient not presenting with ALK gene rearrangement or ROS1 gene rearrangement
* Patient not available for follow-up throughout the duration of the study
* Patient deemed to be incapable of responding to the study questions for linguistic, cognitive or organisational reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with ALK positive or ROS1-positive Locally advanced or metastatic non-small cell lung cancer NSCLC, initiated in the previous 3 months or participants initiating crizotinib treatment regardless of the line of treatment
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- France (26):
  - Centre Hospitalier Intercommunal du Pays d'Aix-Pertuis,Service de Pneumologie, Aix-en-Provence
  - Clinique de l Europe, Amiens
  - Hopital Robert Ballanger, Service de Pneumologie, Aulnay-sous-Bois
  - Centre Hospitalier d Avignon, Avignon
  - Centre Hospitalier de Beauvais, Beauvais
  - Centre Hospitalier General Beziers, Service De Pneumologie, Béziers
  - Centre Hospitalier de Cannes, Cannes
  - Centre Hospitalier Chalon sur Saone William Morey, Chalon-sur-Saône
  - Centre Hospitalier Metropole de Savoie-Site de Chambery, Chambéry
  - Hopitaux Civils de Colmar - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier ALPES LEMAN, Contamine-sur-Arve
  - Centre Hospitalier Intercommunal Frejus, Fréjus
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - CHD Vendee, La Roche-sur-Yon
  - Le Mans Hospital Center, Le Mans
  - Centre Hospitalier des Deux Vallees - Longjumeau BP 125, Longjumeau
  - Hopital Europeen - Service de Pneumologie, Marseille
  - Centre Hospitalier de Macon, Mâcon
  - GHR Mulhouse Sud Alsace, Mulhouse
  - Centre Hospitalier de l'Agglomeration de Nevers, Nevers
  - Centre Hospitalier Regional d Orleans, Orléans
  - Centre Hospitalier Annecy Genevois, Pringy
  - Groupe Hospitalier Sud Reunion, Saint Pierre La Réunion
  - Hopitaux du Leman, Thonon-les-Bains
  - Centre Hospitalier de Troyes, Service de Pneumologie - Oncologie Thoracique, Troyes
  - Centre Hospitalier de Villefranche sur Saone - BP80436, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A8081060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged above or equal to (>=) 18 years, treated with crizotinib for advanced (stage IIIB not suitable for radiotherapy) or metastatic (stage IV) non-small-cell lung cancer (NSCLC), with anaplastic lymphoma kinase-positive (ALK) gene rearrangement or proto-oncogene 1, receptor tyrosine kinase-positive (ROS1) gene rearrangement were observed.
Pre-assignment Details: Participants received crizotinib 3 months before inclusion in the study or initiated crizotinib treatment (regardless of the line of treatment) in general hospitals as per normal routine healthcare practice in real world. Participants were followed up in this observational study for maximum of 18 months post inclusion in the study.
Groups:
- Participants With ALK Gene Rearrangement: Participants included in this arm were treated with crizotinib for advanced or metastatic NSCLC with ALK gene rearrangement, per normal routine medical care in real world practices. The participants were followed from inclusion in the study until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
- Participants With ROS1 Gene Rearrangement: Participants included in this arm were treated with crizotinib for advanced or metastatic NSCLC with ROS1 gene rearrangement, per normal routine medical care in real world practices. The participants were followed from inclusion in the study until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
- Participants With Unknown Gene Rearrangement: Participants included in this arm were treated with crizotinib for advanced or metastatic NSCLC with unknown gene rearrangement, per normal routine medical care in real world practices. The participants were followed from inclusion in the study until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
Period: Overall Study
Arm/Group | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement | Participants With Unknown Gene Rearrangement
Started | 51 | 20 | 2
Safety Population | 51 | 20 | 2
Participants With Known Gene Arrangement; Had First Line Crizotinib | 33 | 18 | 0
Participants With Known Gene Arrangement; Had Second Line Crizotinib | 14 | 1 | 0
Participants With Known Gene Arrangement; Had Third Line Crizotinib | 2 | 0 | 0
Participants With Known Gene Arrangement; Had Other Line Crizotinib | 2 | 1 | 0
Completed | 37 | 8 | 0
Not Completed | 14 | 12 | 2
Not completed — Death | 12 | 11 | 0
Not completed — Other | 0 | 1 | 0
Not completed — Withdrawn due to adverse event (AE) | 2 | 0 | 0
Not completed — Participant not met eligibility criteria | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Participants With ALK Gene Rearrangement: Participants included in this arm were treated with crizotinib for advanced or metastatic NSCLC with ALK gene rearrangement, per normal routine medical care in real world practices. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
- Participants With ROS1 Gene Rearrangement: Participants included in this arm were treated with crizotinib for advanced or metastatic NSCLC with ROS1 gene rearrangement, per normal routine medical care in real world practices. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
- Total: Total of all reporting groups
Arm/Group | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement | Participants With Unknown Gene Rearrangement | Total
Number analyzed (Participants) | 51 | 20 | 2 | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Number analyzed: signify number of participants with evaluable non-missing data.
  Years
    number analyzed (Participants) | 51 | 20 | 1 | 72
    (all) | 60.4 (13.5) | 67.6 (14.4) | 64.0 (NA) — Only 1 participant evaluable, hence standard deviation not estimable. | 62.4 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed: signify number of participants with evaluable non-missing data.
  Participants
    number analyzed (Participants) | 51 | 20 | 1 | 72
    Female | 30 | 15 | 1 | 46
    Male | 21 | 5 | 0 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Age: Line of Treatment
Time Frame: Baseline
Population: FAS included all eligible participants (with known ALK or ROS1 gene rearrangement) who received at least 1 dose of Crizotinib.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Crizotinib: First Line of Treatment: Participants included in this arm were treated with crizotinib as first line of treatment for advanced or metastatic NSCLC with ALK or ROS gene rearrangement, per normal routine medical care in real world practices. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
- Crizotinib: Second Line of Treatment: Participants included in this arm were treated with crizotinib as second line of treatment for advanced or metastatic NSCLC with ALK or ROS gene rearrangement, per normal routine medical care in real world practices. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
- Crizotinib: Third Line of Treatment: Participants included in this arm were treated with crizotinib as third line of treatment for advanced or metastatic NSCLC with ALK or ROS gene rearrangement, per normal routine medical care in real world practices. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
- Crizotinib: Other Line of Treatment: Participants included in this arm were treated with crizotinib as other line than first, second or third of treatment for advanced or metastatic NSCLC with ALK or ROS gene rearrangement, per normal routine medical care in real world practices. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment
Number analyzed (Participants) | 51 | 15 | 2 | 3
Years | 62.3 (15.1) | 63.1 (12.9) | 56.5 (3.5) | 64.3 (3.2)

2. Primary Outcome: Body Weight: Line of Treatment and Gene Rearrangement
Description: Body weight in kilograms (kg) measured at baseline were reported.
Time Frame: Baseline
Population: FAS included all eligible participants (with known ALK or ROS1 gene rearrangement) who received at least 1 dose of Crizotinib. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 14 | 2 | 2 | 49 | 20
Kilogram | 66.5 (15.5) | 69.3 (13.8) | 75.0 (0.0) | 58.5 (14.8) | 69.6 (14.6) | 61.1 (14.1)

3. Primary Outcome: Body Mass Index (BMI): Line of Treatment and Gene Rearrangement
Description: BMI was obtained by dividing body weight in kilograms (kg) by height in meters square (m^2).
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilogram per square meter
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 14 | 2 | 2 | 49 | 20
Kilogram per square meter | 24.34 (4.46) | 24.73 (4.84) | 25.05 (0.78) | 23.50 (4.95) | 25.07 (4.59) | 22.81 (3.57)

4. Primary Outcome: Gender: Line of Treatment
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment
Number analyzed (Participants) | 51 | 15 | 2 | 3
Participants
  Male | 17 | 7 | 2 | 0
  Female | 34 | 8 | 0 | 3

5. Primary Outcome: Number of Participants Classified According to Smoking Status at Baseline: Line of Treatment and Gene Rearrangement
Description: Number of participants were classified according to smoking status as non-smoker, ex-smoker (did not smoke in at least 1 year prior to baseline) and current-smoker.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  Non-smoker | 31 | 7 | 1 | 1 | 28 | 12
  Ex-smoker | 19 | 5 | 1 | 2 | 19 | 8
  Current smoker | 1 | 3 | 0 | 0 | 4 | 0

6. Primary Outcome: Number of Pack Years: Line of Treatment and Gene Rearrangement
Description: The number of pack-years was calculated at baseline for ex-smokers and current smokers by multiplying the number of packs they consumed per day and the number of years that the participant had smoked this quantity of packs. Combined data is reported for ex-smokers and current smokers.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Pack-years
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 20 | 6 | 1 | 2 | 21 | 8
Pack-years | 19.7 (17.2) | 24.5 (9.7) | 60.0 | 10.0 (0.0) | 21.7 (16.1) | 20.5 (19.9)

7. Primary Outcome: Duration of Smoking and Duration of Quitting Smoke: Line of Treatment and Gene Rearrangement
Description: Duration of smoking: a) for ex-smokers, duration of smoking (years) was calculated by subtracting start year with year of smoking stop, b) for current smokers, duration of smoking (years) was calculated by subtracting start year with year of Inclusion visit date. Combined data of duration of smoking is reported for ex-smokers and current smokers. Duration of quitting smoke (years) for ex-smokers was calculated by subtracting year of smoking stop with year of inclusion visit date.
Time Frame: Baseline
Population: FAS included all eligible participants (with known ALK or ROS1 gene rearrangement) who received at least 1 dose of Crizotinib. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows with non-missing data.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 17 | 5 | 1 | 2 | 17 | 8
Years
  Duration of smoking for ex-smokers and current smokers: number analyzed (Participants) | 15 | 5 | 1 | 0 | 14 | 7
  Duration of smoking for ex-smokers and current smokers | 22.6 (13.6) | 26.0 (13.5) | 36.0 |  | 23.1 (12.8) | 25.9 (14.9)
  Duration of quitting smoke for ex-smoker | 12.8 (14.3) | 12.6 (15.4) | 3.0 | 8.0 (2.8) | 10.5 (14.4) | 15.1 (11.6)

8. Primary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Assessment: Line of Treatment and Gene Rearrangement
Description: Number of participants were categorized as yes or no, according to have undergone assessment with ECOG performance status. ECOG performance status was used to measure quality of life of oncology participants with scores running from 0 (no severity) to 5 (maximum severity); where 0= fully active, able to carry on all pre-disease performance without restriction; 1= restricted in physically strenuous activity, ambulatory, able to carry out light or sedentary work; 2= ambulatory, capable of all self-care, unable to carry out any work activity, up greater than (>) 50 percent (%) of waking hours; 3= capable of only limited self-care, confined to bed or chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5= dead.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  No | 5 | 2 | 0 | 1 | 7 | 1
  Yes | 46 | 13 | 2 | 2 | 44 | 19

9. Primary Outcome: Number of Participants Categorized According to ECOG Performance Status Scores: Line of Treatment and Gene Rearrangement
Description: ECOG performance status was used to measure quality of life of oncology patients with scores running from 0 (no severity) to 5 (maximum severity); where 0= fully active, able to carry on all pre-disease performance without restriction; 1= restricted in physically strenuous activity, ambulatory, able to carry out light or sedentary work; 2= ambulatory, capable of all self-care, unable to carry out any work activity, up >50% of waking hours; 3= capable of only limited self-care, confined to bed or chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5= dead. Participants were categorized according to ECOG performance status scores of 0-1 and >=2.
Time Frame: Baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 46 | 13 | 2 | 2 | 44 | 19
Participants
  0-1 | 36 | 12 | 2 | 2 | 38 | 14
  >= 2 | 10 | 1 | 0 | 0 | 6 | 5

10. Primary Outcome: Time Since Diagnosis of NSCLC: Treatment and Gene Rearrangement
Description: Time since diagnosis of NSCLC (months) was calculated as: inclusion visit date minus date of the biopsy that enabled making the diagnosis divided by 365.35/12. If the day of the diagnosis was missing, it was replaced by the 15th of the month for calculation.
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Months | 1.30 [0.70 to 2.30] | 8.00 [3.40 to 39.70] | 48.40 [33.60 to 63.20] | 61.70 [11.70 to 135.90] | 2.70 [1.00 to 6.00] | 1.25 [0.80 to 1.90]

11. Primary Outcome: Number of Participants Categorized According to Type of Tumor's Histology: Line of Treatment and Gene Rearrangement
Description: Participants were categorized according to type of tumor's histology as adenocarcinoma, carcinoma indifferencier and other.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  Adenocarcinoma | 50 | 15 | 2 | 3 | 51 | 19
  Carcinom indifferencier | 1 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 1

12. Primary Outcome: Number of Participants Categorized According to Tumor Stage: Line of Treatment and Gene Rearrangement
Description: Participants were categorized according to tumor stage as IIIA/B or IVA/B classified as per Tumor Node Metastasis (TNM), 8th edition. TNM: based on tumor size, if cancer cells had spread to nearby lymph nodes (LN), or distant (other parts of body) metastasis. Stages included: stage 0 (no evidence of cancer cells), stage l (T1N0M0), stage IIA (T0N1M0, T1N1M0, T2N0M0), stage IIB (T2N1M0, T3N0M0), stage IIIA (T0N2M0, T1N2M0, T2N3M0, T3N1 or N2M0), stage IIIb (T4 any NM0, any TN3M0), stage IIIC (any TN3M0), stage IV (any T any NM1), where T0= early form of tumor, T1=<2 centimeter (cm), T2 =2-5 cm, T3=>2 cm, T4=large sized, N0= not spread to LN, N1= spread to 1 to 3, N2= spread to 4 to 9, N3= spread >10 axillary LN, M0= no metastasis, M1= metastasis. Tumor stage categories with at least 1 participant in any reporting arm are reported.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  IIIA | 0 | 4 | 0 | 0 | 4 | 0
  IIIB | 5 | 0 | 0 | 0 | 3 | 2
  IVA | 18 | 5 | 2 | 1 | 20 | 6
  IVB | 28 | 6 | 0 | 2 | 24 | 12

13. Primary Outcome: Number of Participants Categorized According to Tumor Location: Line of Treatment and Gene Rearrangement
Description: Participants were categorized according to location of tumor: upper right lobe, upper left lobe, middle right lobe, lower right lobe, and lower left lobe.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  Upper right lobe | 15 | 2 | 1 | 1 | 11 | 8
  Upper left lobe | 10 | 6 | 0 | 0 | 12 | 4
  Middle right lobe | 8 | 4 | 0 | 1 | 11 | 2
  Lower right lobe | 9 | 3 | 1 | 0 | 10 | 3
  Lower left lobe | 9 | 0 | 0 | 1 | 7 | 3

14. Primary Outcome: Number of Participants Categorized According to Presence of Metastases: Line of Treatment and Gene Rearrangement
Description: Participants were categorized according to presence of metastases as Yes or No.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  No | 6 | 2 | 0 | 0 | 6 | 2
  Yes | 45 | 13 | 2 | 3 | 45 | 18

15. Primary Outcome: Number of Participants Categorized According to Number of Metastatic Sites: Line of Treatment and Gene Rearrangement
Description: Participants were categorized according to number of metastatic sites.
Time Frame: Baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 45 | 13 | 2 | 3 | 45 | 18
Participants
  1 | 20 | 5 | 1 | 2 | 19 | 9
  2 | 8 | 4 | 1 | 1 | 11 | 3
  >=3 | 17 | 4 | 0 | 0 | 15 | 6

16. Primary Outcome: Number of Participants Categorized According to Location of Metastases: Line of Treatment and Gene Rearrangement
Description: Participants were categorized according to the location of metastases. Participant could have more than 1 location of metastases.
Time Frame: Baseline
Population: FAS included all eligible participants (with known ALK or ROS1 gene rearrangement) who received at least 1 dose of Crizotinib. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 45 | 13 | 2 | 3 | 45 | 18
Participants
  Contralateral lung | 17 | 4 | 1 | 1 | 18 | 5
  Extrathoracic lymph node | 21 | 4 | 1 | 0 | 19 | 7
  Brain | 7 | 1 | 0 | 0 | 7 | 1
  Liver | 9 | 4 | 0 | 0 | 9 | 4
  Bone | 19 | 7 | 1 | 2 | 22 | 7
  Adrenal glands | 2 | 1 | 0 | 0 | 3 | 0
  Pleural effusion | 16 | 4 | 0 | 0 | 12 | 8
  Other | 5 | 0 | 0 | 1 | 3 | 3

17. Primary Outcome: Time Since the First Strategy Start to Crizotinib Initiation: Line of Treatment and Gene Rearrangement
Description: Time since the first strategy start to crizotinib initiation (months) was calculated as: crizotinib initiation date minus start date of the first strategy divided by 365.35/12. If the start date was missing, it was replaced by the 15th of the month for calculation.
Time Frame: Baseline
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 5 | 15 | 2 | 3 | 23 | 2
Months | 1.00 [1.00 to 4.70] | 6.90 [1.10 to 38.70] | 44.45 [29.50 to 59.40] | 60.10 [11.30 to 134.90] | 6.90 [1.00 to 31.70] | 65.95 [60.10 to 71.80]

18. Primary Outcome: Number of Participants Categorized as "Yes" or "No" for Different Lines of Previous Chemotherapy: Line of Treatment and Gene Rearrangement
Description: Number of participants were categorized according to the different lines of chemotherapy.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  First line: Missing | 9 | 0 | 0 | 0 | 4 | 5
  First line: No | 42 | 0 | 0 | 0 | 29 | 13
  First line: Yes | 0 | 15 | 2 | 3 | 18 | 2
  Second line: Missing | 9 | 0 | 0 | 0 | 4 | 5
  Second line: No | 42 | 15 | 0 | 0 | 43 | 14
  Second line: Yes | 0 | 0 | 2 | 3 | 4 | 1
  Third line: Missing | 9 | 0 | 0 | 0 | 4 | 5
  Third line: No | 42 | 15 | 2 | 0 | 45 | 14
  Third line: Yes | 0 | 0 | 0 | 3 | 2 | 1

19. Primary Outcome: Number of Cycles for Different Lines of Previous Chemotherapy: Line of Treatment and Gene Rearrangement
Description: In this outcome measure, median of number of cycles for different lines of chemotherapy were reported.
Time Frame: Baseline
Population: FAS included all eligible participants (with known ALK or ROS1 gene rearrangement) who received at least 1 dose of Crizotinib. "Overall Number of Participants Analyzed" = 0, signifies there were no participants with previous chemotherapy in the respective arms. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows.
Measure: Median (Inter-Quartile Range); unit: Cycles
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 0 | 15 | 2 | 3 | 18 | 2
Cycles
  First line chemotherapy |  | 4.0 [2.0 to 14.0] | 5.0 [4.0 to 6.0] | 4.0 [4.0 to 13.0] | 4.0 [3.0 to 9.0] | 13.5 [13.0 to 14.0]
  Second line chemotherapy: number analyzed (Participants) | 0 | 0 | 2 | 3 | 4 | 1
  Second line chemotherapy |  |  | 3.0 [2.0 to 4.0] | 4.0 [2.0 to 17.0] | 3.0 [2.0 to 4.0] | 17.0 [17.0 to 17.0]
  Third line chemotherapy: number analyzed (Participants) | 0 | 0 | 0 | 3 | 2 | 1
  Third line chemotherapy |  |  |  | 4.0 [1.0 to 27.0] | 14.0 [1.0 to 27.0] | 4.0 [4.0 to 4.0]

20. Primary Outcome: Duration of Different Lines of Previous Chemotherapy: Line of Treatment and Gene Rearrangement
Description: In this outcome measure, median duration of different lines of chemotherapy was reported. Duration of chemotherapy (months) was calculated as = End date of the last cycle minus start date of the first cycle plus 1 divided by 365.25/12. If the day of the date was missing, it was replaced by the 15th of the month. If the month of the date was missing, the duration was considered as missing.
Time Frame: Baseline
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 0 | 15 | 2 | 3 | 18 | 2
Months
  First line chemotherapy |  | 2.70 [0.80 to 9.00] | 3.60 [2.10 to 5.10] | 2.60 [0.70 to 11.90] | 2.65 [0.80 to 6.30] | 11.30 [10.70 to 11.90]
  Second line chemotherapy: number analyzed (Participants) | 0 | 0 | 2 | 3 | 4 | 1
  Second line chemotherapy |  |  | 1.85 [1.10 to 2.60] | 1.30 [0.70 to 2.10] | 1.20 [0.90 to 1.95] | 2.10 [2.10 to 2.10]
  Third line chemotherapy: number analyzed (Participants) | 0 | 0 | 0 | 3 | 2 | 1
  Third line chemotherapy |  |  |  | 3.30 [0.50 to 41.80] | 21.15 [0.50 to 41.80] | 3.30 [3.30 to 3.30]

21. Primary Outcome: Number of Participants Categorized as "Yes" or "No" for Previous Brain Irradiation Therapy, Previous Radiotherapies and Previous Tyrosine Kinase Inhibitor Therapy: Line of Treatment and Gene Rearrangement
Description: In this outcome measure, participants were categorized according to the previous treatments received. Participant could have received more than 1 type of previous therapies.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  Brain irradiation: Missing | 6 | 0 | 0 | 0 | 2 | 4
  Brain irradiation: No | 44 | 15 | 2 | 3 | 48 | 16
  Brain irradiation: Yes | 1 | 0 | 0 | 0 | 1 | 0
  Radiotherapies: Missing | 5 | 0 | 0 | 0 | 2 | 3
  Radiotherapies: No | 44 | 11 | 2 | 0 | 42 | 15
  Radiotherapies: Yes | 2 | 4 | 0 | 3 | 7 | 2
  Tyrosine Kinase inhibitor: Missing | 0 | 0 | 0 | 0 | 0 | 0
  Tyrosine Kinase inhibitor: No | 51 | 15 | 2 | 3 | 51 | 20
  Tyrosine Kinase inhibitor: Yes | 0 | 0 | 0 | 0 | 0 | 0

22. Primary Outcome: Dose of Previous Brain Irradiation and Radiotherapies: Line of Treatment and Gene Rearrangement
Description: In this outcome measure, median of dose of brain irradiation and radiotherapies were reported.
Time Frame: Baseline
Population: FAS included all eligible participants (with known ALK or ROS1 gene rearrangement) who received at least 1 dose of Crizotinib. "Overall Number of Participants Analyzed" = 0, signifies there were no participants with brain irradiation therapy and radiotherapy in respective arms. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows.
Measure: Median (Inter-Quartile Range); unit: Gray unit
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 2 | 4 | 0 | 3 | 7 | 2
Gray unit
  Brain irradiation dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0
  Brain irradiation dose | 30.0 [30.0 to 30.0] |  |  |  | 30.0 [30.0 to 30.0] |
  Radiotherapy dose | 20.0 [20.0 to 20.0] | 42.5 [30.0 to 57.0] |  | 30.0 [30.0 to 30.0] | 30.0 [30.0 to 55.0] | 25.0 [20.0 to 30.0]

23. Primary Outcome: Duration of Previous Brain Irradiation Therapy and Radiotherapies: Line of Treatment and Gene Rearrangement
Description: In this outcome measure, duration of previous brain irradiation therapy and radiotherapies was reported.
Time Frame: Baseline
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 2 | 4 | 0 | 3 | 7 | 2
Months
  Brain Irradiation therapy: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0
  Brain Irradiation therapy | 15.0 [15.0 to 15.0] |  |  |  | 15.0 [15.0 to 15.0] |
  Radiotherapies | 7.0 [7.0 to 7.0] | 30.5 [16.0 to 46.5] |  | 15.0 [12.0 to 16.0] | 15.0 [12.0 to 43.0] | 11.5 [7.0 to 16.0]

24. Secondary Outcome: Number of Participants Categorized According to Diagnostic Method to Detect ALK and ROS1 Gene Rearrangement: Line of Treatment and Gene Rearrangement
Description: In this outcome measure, the number of participants were categorized according to diagnostic method used to detect ALK and ROS1 gene rearrangement.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  Histology | 47 | 13 | 2 | 2 | 44 | 20
  Cytology | 4 | 2 | 0 | 1 | 7 | 0

25. Secondary Outcome: Number of Participants Categorized According to Origin of Specimen to Detect ALK and ROS1 Gene Rearrangement: Line of Treatment and Gene Rearrangement
Description: In this outcome measure, number of participants were categorized according to origin of specimen to detect ALK and ROS1 gene rearrangement. Origins of specimen included: primitive tumor, thoracic lymph node, extrathoracic lymph node, bone, adrenal glands and pleural.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  Primitive tumor | 37 | 10 | 2 | 3 | 36 | 16
  Thoracic lymph node | 4 | 2 | 0 | 0 | 4 | 2
  Extrathoracic lymph node | 3 | 0 | 0 | 0 | 3 | 0
  Bone | 1 | 0 | 0 | 0 | 1 | 0
  Adrenal glands | 0 | 1 | 0 | 0 | 1 | 0
  Pleural | 6 | 2 | 0 | 0 | 6 | 2

26. Secondary Outcome: Number of Participants Categorized According to Analysis Platform to Detect ALK and ROS1 Gene Rearrangement: Line of Treatment and Gene Rearrangement
Description: In this outcome measure, number of participants were categorized according to analysis platform to detect ALK and ROS1 gene rearrangement. Analysis platform included following sites: University hospital center (UHC) Alsace Cancer center of Strasbourg - Hospital Center of Mulhouse - Hospital Center of Colmar; UHC Aquitaine - Hospital Center de Bordeaux - La Réunion; UHC Bourgogne - Hospital Center of Dijon, UHC of Tours - Orléans; UHC Haute-Normandie - Hospital Center of Rouen, Ile-de-France AP - HP; UHC Languedoc Roussillon - Hospital Center of Montpellier - UHC of Nîmes; UHC Nord-Pas-de-Calais - Hospital Center of Lille; UHC Pays-de-la-Loire - Hospital Center of Nantes; UHC Pays-de-la-Loire - Hospital Center of Angers; UHC Picardie, Amiens; UHC Provence Alpes Côte d'Azur - Hospital Center of Nice; UHC Provence Alpes Côte d'Azur - Hospital Center of Marseille; UHC Rhône Alpes - Hospital Center of Lyon; UHC Rhône Alpes - Hospital Center of Grenoble; and other platform.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  UHC Alsace Cancer center of Strasbourg - Hospital Center of Mulhouse - Hospital Center of Colmar | 10 | 1 | 0 | 0 | 4 | 7
  UHC Aquitaine - Hospital Center de Bordeaux - La Réunion | 1 | 0 | 0 | 0 | 1 | 0
  UHC Bourgogne - Hospital Center of Dijon | 0 | 2 | 0 | 1 | 3 | 0
  UHC of Tours - Orléans | 6 | 1 | 0 | 0 | 6 | 1
  UHC Haute-Normandie - Hospital Center of Rouen | 0 | 1 | 0 | 0 | 1 | 0
  Ile-de-France AP - HP | 2 | 0 | 1 | 0 | 3 | 0
  UHC Languedoc Roussillon - Hospital Center of Montpellier - University hospital center of Nîmes | 2 | 0 | 1 | 0 | 3 | 0
  UHC Nord-Pas-de-Calais - Hospital Center of Lille | 1 | 0 | 0 | 0 | 1 | 0
  UHC Pays-de-la-Loire - Hospital Center of Nantes | 4 | 0 | 0 | 0 | 2 | 2
  UHC Pays-de-la-Loire - Hospital Center of Angers | 3 | 1 | 0 | 1 | 5 | 0
  UHC Picardie, Amiens | 1 | 0 | 0 | 0 | 1 | 0
  UHC Provence Alpes Côte d'Azur - Hospital Center of Nice | 3 | 0 | 0 | 0 | 3 | 0
  UHC Provence Alpes Côte d'Azur - Hospital Center of Marseille | 0 | 1 | 0 | 0 | 1 | 0
  UHC Rhône Alpes - Hospital Center of Lyon | 2 | 2 | 0 | 1 | 3 | 2
  UHC Rhône Alpes - Hospital Center of Grenoble | 8 | 5 | 0 | 0 | 9 | 4
  Other platform | 8 | 1 | 0 | 0 | 5 | 4

27. Secondary Outcome: Number of Participants Categorized According to Technique Used to Detect ALK and ROS1 Gene Rearrangement: Line of Treatment and Gene Rearrangement
Description: In this outcome measure, number of participants were categorized according to the techniques used to detect ALK and ROS1 gene rearrangement. Techniques involved were: Immunohistochemistry (IHC); Fluorescence in situ hybridisation (FISH); Reverse transcriptase polymerase chain reaction (RT-PCR); Next-Generation Sequencing (NGS); Other; and Associations-FISH, IHC, IHC+FISH, IHC+FISH+NGS, NGS.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  IHC | 46 | 14 | 2 | 2 | 47 | 17
  FISH | 34 | 12 | 2 | 1 | 32 | 17
  RT-PCR | 0 | 0 | 0 | 0 | 0 | 0
  NGS | 16 | 2 | 1 | 0 | 12 | 7
  Other | 0 | 0 | 0 | 0 | 0 | 0
  Associations: FISH | 4 | 1 | 0 | 1 | 3 | 3
  Associations: IHC | 14 | 2 | 0 | 2 | 15 | 3
  Associations: IHC+FISH | 17 | 10 | 1 | 0 | 21 | 7
  Associations: IHC+FISH+NGS | 13 | 1 | 1 | 0 | 8 | 7
  Associations: IHC+NGS | 2 | 1 | 0 | 0 | 3 | 0
  Associations: NGS | 1 | 0 | 0 | 0 | 1 | 0

28. Secondary Outcome: Duration Between Sending and Receipt of ALK and ROS1 Results: Line of Treatment and Gene Rearrangement
Description: Duration between sending and receipt of ALK for positive ALK was calculated in days by subtracting the date sent to the platform from date when positive ALK result was received. Duration between sending and receipt of ROS1 for positive ROS1 was calculated in days by subtracting the date sent to the platform from date when positive ROS1 result was received.
Time Frame: Baseline
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 33 | 14 | 2 | 2 | 51 | 20
Days
  ALK+: number analyzed (Participants) | 33 | 14 | 2 | 2 | 51 | 0
  ALK+ | 8.0 [3.0 to 14.0] | 18.0 [10.0 to 26.0] | 19.5 [19.0 to 20.0] | 11.0 [3.0 to 19.0] | 10.0 [4.0 to 19.0] |
  ROS1+: number analyzed (Participants) | 18 | 1 | 0 | 1 | 0 | 20
  ROS1+ | 8.0 [7.0 to 13.0] | 5.0 [5.0 to 5.0] |  | 8.0 [8.0 to 8.0] |  | 8.0 [6.5 to 12.5]

29. Secondary Outcome: Number of Participants Among Whom Search for Other Biological Markers Was Carried Out: Line of Treatment and Gene Rearrangement
Description: In this outcome measure, number of participants were categorized "Yes" or "No" for search of other biological markers.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Participants
  No | 2 | 4 | 0 | 0 | 4 | 2
  Yes | 49 | 11 | 2 | 3 | 47 | 18

30. Secondary Outcome: Number of Participants Categorized According to Clinical Response at Month 3, 6, 9, 12, 15 and 18
Description: Number of participants were categorized according to clinical response as evaluated by physician. Clinical response was categorized into disease improvement, disease stabilization or disease degradation.
Time Frame: Month 3, 6, 9, 12, 15 and 18
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Groups:
- Crizotinib: ALK+ NSCLC: Participants aged >=18 years, followed up for locally advanced (stage IIIB not suitable for radiotherapy) or metastatic (stage IV) ALK+ NSCLC initiating (or having initiated in previous 3 months) treatment with crizotinib regardless of the line of treatment were sequentially included in this observational, descriptive, longitudinal, multicentre, retro-prospective study. The participants received crizotinib as per normal routine healthcare practice in real world. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
- Crizotinib: ROS+ NSCLC: Participants aged >=18 years, followed up for locally advanced (stage IIIB not suitable for radiotherapy) or metastatic (stage IV) ALK+ NSCLC initiating (or having initiated in previous 3 months) treatment with crizotinib regardless of line of treatment were sequentially included in this observational, descriptive, longitudinal, multicentre, retro-prospective study. The participants received crizotinib as per normal routine healthcare practice in real world. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 48 | 14 | 2 | 3 | 48 | 19
Participants
  Month 3: Missing | 0 | 0 | 0 | 0 | 0 | 0
  Month 3: Improvement | 21 | 6 | 1 | 3 | 21 | 10
  Month 3: Disease stabilization | 20 | 8 | 0 | 0 | 22 | 6
  Month 3: Disease degradation | 7 | 0 | 1 | 0 | 5 | 3
  Month 6: number analyzed (Participants) | 38 | 12 | 1 | 3 | 40 | 14
  Month 6: Missing | 0 | 0 | 0 | 0 | 0 | 0
  Month 6: Improvement | 14 | 2 | 0 | 1 | 13 | 4
  Month 6: Disease stabilization | 17 | 7 | 1 | 0 | 18 | 7
  Month 6: Disease degradation | 7 | 3 | 0 | 2 | 9 | 3
  Month 9: number analyzed (Participants) | 29 | 7 | 1 | 1 | 28 | 10
  Month 9: Missing | 0 | 0 | 0 | 0 | 0 | 0
  Month 9: Improvement | 9 | 1 | 0 | 0 | 8 | 2
  Month 9: Disease stabilization | 18 | 5 | 1 | 0 | 17 | 7
  Month 9: Disease degradation | 2 | 1 | 0 | 1 | 3 | 1
  Month 12: number analyzed (Participants) | 24 | 7 | 1 | 1 | 26 | 7
  Month 12: Missing | 0 | 1 | 0 | 0 | 1 | 0
  Month 12: Improvement | 6 | 1 | 0 | 0 | 5 | 2
  Month 12: Disease stabilization | 17 | 5 | 1 | 1 | 20 | 4
  Month 12: Disease degradation | 1 | 0 | 0 | 0 | 0 | 1
  Month 15: number analyzed (Participants) | 17 | 7 | 1 | 0 | 22 | 3
  Month 15: Missing | 0 | 1 | 0 |  | 1 | 0
  Month 15: Improvement | 2 | 0 | 0 |  | 1 | 1
  Month 15: Disease stabilization | 12 | 6 | 1 |  | 18 | 1
  Month 15: Disease degradation | 3 | 0 | 0 |  | 2 | 1
  Month 18: number analyzed (Participants) | 16 | 5 | 1 | 0 | 18 | 4
  Month 18: Missing | 1 | 0 | 0 |  | 0 | 1
  Month 18: Improvement | 1 | 0 | 0 |  | 0 | 1
  Month 18: Disease stabilization | 14 | 5 | 1 |  | 18 | 2
  Month 18: Disease degradation | 0 | 0 | 0 |  | 0 | 0

31. Secondary Outcome: Number of Participants Categorized According to Tumor Response at Month 3, 6, 9, 12, 15 and 18
Description: Number of participants were categorized according to tumor response per Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. Tumor response included total (complete) response (CR), partial response (PR), stable disease (SD) or disease progression (PD) on imaging. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Persistence of one or more non-target lesion and/or maintenance of tumor marker level above the normal limits. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. Unequivocal progression of existing non-target lesions. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Month 3, 6, 9, 12, 15 and 18
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 48 | 14 | 2 | 3 | 48 | 19
Participants
  Month 3: Missing | 4 | 0 | 0 | 0 | 1 | 3
  Month 3: Total response | 1 | 2 | 0 | 0 | 1 | 2
  Month 3: Partial response | 25 | 6 | 1 | 2 | 27 | 7
  Month 3: Disease stable | 13 | 4 | 0 | 1 | 12 | 6
  Month 3: Progression | 5 | 2 | 1 | 0 | 7 | 1
  Month 6: number analyzed (Participants) | 38 | 12 | 1 | 3 | 40 | 14
  Month 6: Missing | 0 | 0 | 0 | 0 | 0 | 0
  Month 6: Total response | 1 | 1 | 0 | 0 | 0 | 2
  Month 6: Partial response | 19 | 4 | 1 | 1 | 22 | 3
  Month 6: Disease stable | 7 | 3 | 0 | 1 | 7 | 4
  Month 6: Progression | 11 | 4 | 0 | 1 | 11 | 5
  Month 9: number analyzed (Participants) | 29 | 7 | 1 | 1 | 28 | 10
  Month 9: Missing | 0 | 0 | 0 | 0 | 0 | 0
  Month 9: Total response | 2 | 1 | 0 | 0 | 0 | 3
  Month 9: Partial response | 16 | 3 | 1 | 0 | 18 | 2
  Month 9: Disease stable | 6 | 2 | 0 | 1 | 6 | 3
  Month 9: Progression | 5 | 1 | 0 | 0 | 4 | 2
  Month 12: number analyzed (Participants) | 24 | 7 | 1 | 1 | 26 | 7
  Month 12: Missing | 0 | 1 | 0 | 0 | 1 | 0
  Month 12: Total response | 1 | 2 | 0 | 0 | 2 | 1
  Month 12: Partial response | 14 | 2 | 1 | 1 | 14 | 4
  Month 12: Disease stable | 5 | 1 | 0 | 0 | 5 | 1
  Month 12: Progression | 4 | 1 | 0 | 0 | 4 | 1
  Month 15: number analyzed (Participants) | 17 | 7 | 1 | 0 | 22 | 3
  Month 15: Missing | 0 | 1 | 0 |  | 1 | 0
  Month 15: Total response | 1 | 2 | 0 |  | 2 | 1
  Month 15: Partial response | 8 | 1 | 1 |  | 9 | 1
  Month 15: Disease stable | 3 | 2 | 0 |  | 5 | 0
  Month 15: Progression | 5 | 1 | 0 | 0 | 5 | 1
  Month 18: number analyzed (Participants) | 16 | 5 | 1 | 0 | 18 | 4
  Month 18: Missing | 1 | 0 | 0 |  | 0 | 1
  Month 18: Total response | 1 | 2 | 0 |  | 2 | 1
  Month 18: Partial response | 9 | 1 | 1 |  | 10 | 1
  Month 18: Disease stable | 5 | 1 | 0 |  | 5 | 1
  Month 18: Progression | 0 | 1 | 0 |  | 1 | 0

32. Secondary Outcome: Time Since Diagnosis to Progression at Month 3, 6, 9, 12, 15 and 18
Description: Time since diagnosis to progression (months) was calculated as: progression date minus date of biopsy that enabled making the diagnosis divided by 365.35/12. If the day of the diagnosis was missing, it was replaced by the 15th of the month for calculation. If the day of the progression was missing, it was replaced by the 1st of the month for calculation.
Time Frame: Month 3, 6, 9, 12, 15 and 18
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 11 | 4 | 1 | 1 | 11 | 5
Months
  Month 3: number analyzed (Participants) | 5 | 2 | 1 | 0 | 7 | 1
  Month 3 | 4.30 [3.00 to 6.60] | 35.45 [15.20 to 55.70] | 35.90 [35.90 to 35.90] |  | 6.70 [4.30 to 35.90] | 2.90 [2.90 to 2.90]
  Month 6: number analyzed (Participants) | 11 | 4 | 0 | 1 | 11 | 5
  Month 6 | 7.10 [6.50 to 7.70] | 16.85 [13.50 to 32.05] |  | 140.60 [140.60 to 140.60] | 10.40 [6.50 to 17.50] | 7.30 [7.10 to 7.50]
  Month 9: number analyzed (Participants) | 5 | 1 | 0 | 0 | 4 | 2
  Month 9 | 9.30 [8.70 to 11.70] | 62.90 [62.90 to 62.90] |  |  | 10.50 [8.25 to 37.30] | 10.30 [8.70 to 11.90]
  Month 12: number analyzed (Participants) | 4 | 1 | 0 | 0 | 4 | 1
  Month 12 | 11.35 [10.40 to 12.35] | 50.60 [50.60 to 50.60] |  |  | 11.35 [10.40 to 31.25] | 12.80 [12.80 to 12.80]
  Month 15: number analyzed (Participants) | 5 | 1 | 0 | 0 | 5 | 1
  Month 15 | 17.00 [15.10 to 17.50] | 17.80 [17.80 to 17.80] |  |  | 17.50 [17.00 to 17.80] | 15.10 [15.10 to 15.10]
  Month 18: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0
  Month 18 |  | 57.50 [57.50 to 57.50] |  |  | 57.50 [57.50 to 57.50] |

33. Secondary Outcome: Number of Participants With Site of Progression as Primary Tumor at Month 3, 6, 9, 12, 15 and 18
Description: In this outcome measure, number of participants whose progression was noted at primary tumor site were reported.
Time Frame: Month 3, 6, 9, 12, 15 and 18
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 11 | 4 | 1 | 1 | 11 | 5
Participants
  Month 3: number analyzed (Participants) | 5 | 2 | 1 | 0 | 7 | 1
  Month 3 | 1 | 0 | 1 |  | 1 | 1
  Month 6: number analyzed (Participants) | 11 | 4 | 0 | 1 | 11 | 5
  Month 6 | 2 | 0 |  | 0 | 1 | 1
  Month 9: number analyzed (Participants) | 5 | 1 | 0 | 0 | 4 | 2
  Month 9 | 1 | 1 |  |  | 2 | 0
  Month 12: number analyzed (Participants) | 4 | 1 | 0 | 0 | 4 | 1
  Month 12 | 1 | 1 |  |  | 2 | 0
  Month 15: number analyzed (Participants) | 5 | 1 | 0 | 0 | 5 | 1
  Month 15 | 0 | 1 |  |  | 1 | 0
  Month 18: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0
  Month 18 |  | 0 |  |  | 0 |

34. Secondary Outcome: Number of Participants With Site of Progression as Already Existing Metastasis at Month 3, 6, 9, 12, 15 and 18
Description: In this outcome measure, number of participants whose progression was noted at already existing metastasis sites were reported.
Time Frame: Month 3, 6, 9, 12, 15 and 18
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 11 | 4 | 1 | 1 | 11 | 5
Participants
  Month 3: number analyzed (Participants) | 5 | 2 | 1 | 0 | 7 | 1
  Month 3 | 4 | 2 | 1 |  | 6 | 1
  Month 6: number analyzed (Participants) | 11 | 4 | 0 | 1 | 11 | 5
  Month 6 | 6 | 2 |  | 0 | 4 | 4
  Month 9: number analyzed (Participants) | 5 | 1 | 0 | 0 | 4 | 2
  Month 9 | 4 | 0 |  |  | 2 | 2
  Month 12: number analyzed (Participants) | 4 | 1 | 0 | 0 | 4 | 1
  Month 12 | 2 | 0 |  |  | 1 | 1
  Month 15: number analyzed (Participants) | 5 | 1 | 0 | 0 | 5 | 1
  Month 15 | 3 | 0 |  |  | 2 | 1
  Month 18: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0
  Month 18 |  | 0 |  |  | 0 |

35. Secondary Outcome: Number of Participants Categorized According to Location of Progression in Already Existing Metastasis at Month 3, 6, 9, 12, 15 and 18
Description: In this outcome measure, participants were categorized according to location of progression in already existing metastasis which were located at adrenal glands, bone, brain, liver, lymph node, pleural, plueral liver, pleural lymph node, brain pleural, and kidney. Only those rows are reported with at least 1 participant as data for any reporting arm.
Time Frame: Month 3, 6, 9, 12, 15 and 18
Population: FAS analyzed. "Overall Number of Participants Analyzed" = 0, signifies there was no participant with progression at already existing metastasis sites in respective arm. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows. At Month 18 no participant had progression at already existing metastasis sites for any reporting arm, hence no rows for Month 18 are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 6 | 2 | 1 | 0 | 6 | 4
Participants
  Adrenal glands: Month 3: number analyzed (Participants) | 4 | 2 | 1 | 0 | 6 | 1
  Adrenal glands: Month 3 | 0 | 1 | 0 |  | 1 | 0
  Bone: Month 3: number analyzed (Participants) | 4 | 2 | 1 | 0 | 6 | 1
  Bone: Month 3 | 1 | 0 | 0 |  | 0 | 1
  Brain: Month 3: number analyzed (Participants) | 4 | 2 | 1 | 0 | 6 | 1
  Brain: Month 3 | 2 | 0 | 0 |  | 2 | 0
  Liver: Month 3: number analyzed (Participants) | 4 | 2 | 1 | 0 | 6 | 1
  Liver: Month 3 | 0 | 1 | 0 |  | 1 | 0
  Lymph node: Month 3: number analyzed (Participants) | 4 | 2 | 1 | 0 | 6 | 1
  Lymph node: Month 3 | 0 | 0 | 1 |  | 1 | 0
  Pleural, liver: Month 3: number analyzed (Participants) | 4 | 2 | 1 | 0 | 6 | 1
  Pleural, liver: Month 3 | 1 | 0 | 0 |  | 1 | 0
  Adrenal glands: Month 6: number analyzed (Participants) | 6 | 2 | 0 | 0 | 4 | 4
  Adrenal glands: Month 6 | 0 | 1 |  |  | 1 | 0
  Bone: Month 6: number analyzed (Participants) | 6 | 2 | 0 | 0 | 4 | 4
  Bone: Month 6 | 1 | 0 |  |  | 1 | 0
  Brain: Month 6: number analyzed (Participants) | 6 | 2 | 0 | 0 | 4 | 4
  Brain: Month 6 | 2 | 0 |  |  | 0 | 2
  Lymph node: Month 6: number analyzed (Participants) | 6 | 2 | 0 | 0 | 4 | 4
  Lymph node: Month 6 | 0 | 1 |  |  | 1 | 0
  Pleural: Month 6: number analyzed (Participants) | 6 | 2 | 0 | 0 | 4 | 4
  Pleural: Month 6 | 2 | 0 |  |  | 1 | 1
  Pleural, lymph node: Month 6: number analyzed (Participants) | 6 | 2 | 0 | 0 | 4 | 4
  Pleural, lymph node: Month 6 | 1 | 0 |  |  | 0 | 1
  Brain: Month 9: number analyzed (Participants) | 4 | 0 | 0 | 0 | 2 | 2
  Brain: Month 9 | 1 |  |  |  | 0 | 1
  Brain, pleural: Month 9: number analyzed (Participants) | 4 | 0 | 0 | 0 | 2 | 2
  Brain, pleural: Month 9 | 1 |  |  |  | 1 | 0
  Lymph node: Month 9: number analyzed (Participants) | 4 | 0 | 0 | 0 | 2 | 2
  Lymph node: Month 9 | 1 |  |  |  | 0 | 1
  Other: Month 9: number analyzed (Participants) | 4 | 0 | 0 | 0 | 2 | 2
  Other: Month 9 | 1 |  |  |  | 1 | 0
  Brain: Month 12: number analyzed (Participants) | 2 | 0 | 0 | 0 | 1 | 1
  Brain: Month 12 | 1 |  |  |  | 1 | 0
  Brain, liver, bone: Month 12: number analyzed (Participants) | 2 | 0 | 0 | 0 | 1 | 1
  Brain, liver, bone: Month 12 | 1 |  |  |  | 0 | 1
  Kidney: Month 15: number analyzed (Participants) | 3 | 0 | 0 | 0 | 2 | 1
  Kidney: Month 15 | 1 |  |  |  | 1 | 0
  Liver: Month 15: number analyzed (Participants) | 3 | 0 | 0 | 0 | 2 | 1
  Liver: Month 15 | 1 |  |  |  | 1 | 0
  Lymph node: Month 15: number analyzed (Participants) | 3 | 0 | 0 | 0 | 2 | 1
  Lymph node: Month 15 | 1 |  |  |  | 0 | 1

36. Secondary Outcome: Number of Participants With Site of Progression as New Metastases at Month 3, 6, 9, 12, 15 and 18
Description: In this outcome measure, participants with new metastases as the site of progression were reported.
Time Frame: Month 3, 6, 9, 12, 15 and 18
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 11 | 4 | 1 | 1 | 11 | 5
Participants
  Month 3: number analyzed (Participants) | 5 | 2 | 1 | 0 | 7 | 1
  Month 3 | 3 | 1 | 0 |  | 3 | 1
  Month 6: number analyzed (Participants) | 11 | 4 | 0 | 1 | 11 | 5
  Month 6 | 3 | 3 |  | 1 | 7 | 0
  Month 9: number analyzed (Participants) | 5 | 1 | 0 | 0 | 4 | 2
  Month 9 | 1 | 1 |  |  | 1 | 1
  Month 12: number analyzed (Participants) | 4 | 1 | 0 | 0 | 4 | 1
  Month 12 | 2 | 1 |  |  | 2 | 0
  Month 15: number analyzed (Participants) | 5 | 1 | 0 | 0 | 5 | 1
  Month 15 | 5 | 0 |  |  | 4 | 1
  Month 18: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0
  Month 18 |  | 1 |  |  | 1 |

37. Secondary Outcome: Number of Participants Categorized According to Location of Site of Progression as New Metastases at Month 3, 6, 9, 12, 15 and 18
Description: In this outcome measure, number of participants were categorized according to progression at location of new metastases. Location of new metastases included contralateral lung, extrathoracic lymph node, brain, liver, bone, adrenal glands, lymphangite carcinomateuse and pleural. Only those categories in which at least 1 participant had data were reported.
Time Frame: Month 3, 6, 9, 12, 15 and 18
Population: FAS included all eligible participants (with known ALK or ROS1 gene rearrangement) who received at least 1 dose of Crizotinib. "Overall Number of Participants Analyzed" = 0, signifies there was no participant with new metastases as site of progression in the respective arm. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 5 | 3 | 0 | 1 | 7 | 1
Participants
  Brain: Month 3: number analyzed (Participants) | 3 | 1 | 0 | 0 | 3 | 1
  Brain: Month 3 | 2 | 1 |  |  | 3 | 0
  Bone: Month 3: number analyzed (Participants) | 3 | 1 | 0 | 0 | 3 | 1
  Bone: Month 3 | 1 | 0 |  |  | 0 | 1
  Contralateral lung: Month 6: number analyzed (Participants) | 3 | 3 | 0 | 1 | 7 | 0
  Contralateral lung: Month 6 | 0 | 1 |  | 0 | 1 |
  Extrathoracic lymph node: Month 6: number analyzed (Participants) | 3 | 3 | 0 | 1 | 7 | 0
  Extrathoracic lymph node: Month 6 | 1 | 0 |  | 0 | 1 |
  Brain: Month 6: number analyzed (Participants) | 3 | 3 | 0 | 1 | 7 | 0
  Brain: Month 6 | 3 | 3 |  | 0 | 6 |
  Bone: Month 6: number analyzed (Participants) | 3 | 3 | 0 | 1 | 7 | 0
  Bone: Month 6 | 0 | 1 |  | 0 | 1 |
  Lymphangite carcinomateuse: Month 6: number analyzed (Participants) | 3 | 3 | 0 | 1 | 7 | 0
  Lymphangite carcinomateuse: Month 6 | 0 | 1 |  | 0 | 1 |
  Pleural: Month 6: number analyzed (Participants) | 3 | 3 | 0 | 1 | 7 | 0
  Pleural: Month 6 | 0 | 1 |  | 1 | 2 |
  Extrathoracic lymph node: Month 9: number analyzed (Participants) | 1 | 1 | 0 | 0 | 1 | 1
  Extrathoracic lymph node: Month 9 | 0 | 1 |  |  | 1 | 0
  Brain: Month 9: number analyzed (Participants) | 1 | 1 | 0 | 0 | 1 | 1
  Brain: Month 9 | 1 | 0 |  |  | 0 | 1
  Other: Month 9: number analyzed (Participants) | 1 | 1 | 0 | 0 | 1 | 1
  Other: Month 9 | 0 | 1 |  |  | 1 | 0
  Bone: Month 12: number analyzed (Participants) | 2 | 1 | 0 | 0 | 2 | 0
  Bone: Month 12 | 1 | 0 |  |  | 1 |
  Other: Month 12: number analyzed (Participants) | 2 | 0 | 0 | 0 | 2 | 0
  Other: Month 12 | 1 |  |  |  | 1 |
  Contralateral lung: Month 15: number analyzed (Participants) | 5 | 0 | 0 | 0 | 4 | 1
  Contralateral lung: Month 15 | 2 |  |  |  | 1 | 1
  Extrathoracic lymph node: Month 15: number analyzed (Participants) | 5 | 0 | 0 | 0 | 4 | 1
  Extrathoracic lymph node: Month 15 | 1 |  |  |  | 1 | 0
  Brain: Month 15: number analyzed (Participants) | 5 | 0 | 0 | 0 | 4 | 1
  Brain: Month 15 | 4 |  |  |  | 3 | 1
  Other: Month 15: number analyzed (Participants) | 5 | 0 | 0 | 0 | 4 | 1
  Other: Month 15 | 1 |  |  |  | 1 | 0
  Extrathoracic lymph node: Month 18: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0
  Extrathoracic lymph node: Month 18 |  | 1 |  |  | 1 |

38. Secondary Outcome: Treatment Duration Until Progression With Brain Metastases
Description: Treatment duration until progression with brain metastases (weeks) was calculated as: ([date of progression - first treatment intake date] + 1) divided by 7. If the day of the progression was missing, it was replaced by the 1st of the month for calculation.
Time Frame: Baseline
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 8 | 3 | 0 | 0 | 10 | 1
Months | 35.55 [26.50 to 66.55] | 29.70 [22.00 to 36.30] |  |  | 29.40 [26.10 to 42.00] | 62.00 [62.00 to 62.00]

39. Secondary Outcome: Number of Participants With Biopsy on Progression at Month 3, 6, 9, 12, 15 and 18
Description: In this outcome measure, number of participants were categorized on the basis of conduction of biopsy on progression as "Yes' or "No".
Time Frame: Month 3, 6, 9, 12, 15 and 18
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 11 | 4 | 1 | 1 | 11 | 5
Participants
  Month 3: number analyzed (Participants) | 5 | 2 | 1 | 0 | 7 | 1
  Month 3: No | 4 | 1 | 0 |  | 4 | 1
  Month 3: Yes | 1 | 1 | 1 |  | 3 | 0
  Month 3: Missing | 0 | 0 | 0 |  | 0 | 0
  Month 6: number analyzed (Participants) | 11 | 4 | 0 | 1 | 11 | 5
  Month 6: No | 10 | 4 |  | 0 | 10 | 4
  Month 6: Yes | 1 | 0 |  | 1 | 1 | 1
  Month 6: Missing | 0 | 0 |  | 0 | 0 | 0
  Month 9: number analyzed (Participants) | 5 | 1 | 0 | 0 | 4 | 2
  Month 9: No | 4 | 0 |  |  | 3 | 1
  Month 9: Yes | 1 | 1 |  |  | 1 | 1
  Month 9: Missing | 0 | 0 |  |  | 0 | 0
  Month 12: number analyzed (Participants) | 4 | 1 | 0 | 0 | 4 | 1
  Month 12: No | 4 | 1 |  |  | 4 | 1
  Month 12: Yes | 0 | 0 |  |  | 0 | 0
  Month 12: Missing | 0 | 0 |  |  | 0 | 0
  Month 15: number analyzed (Participants) | 5 | 1 | 0 | 0 | 5 | 1
  Month 15: No | 4 | 1 |  |  | 5 | 0
  Month 15: Yes | 0 | 0 |  |  | 0 | 0
  Month 15: Missing | 1 | 0 |  |  | 0 | 1
  Month 18: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0
  Month 18: No |  | 1 |  |  | 1 |
  Month 18: Yes |  | 0 |  |  | 0 |
  Month 18: Missing |  | 0 |  |  | 0 |

40. Secondary Outcome: Objective Response Rate (ORR)
Description: The objective response rate was defined as the percentage of participants with complete response (CR) or partial response (PR) based on RECIST v1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Persistence of one or more non-target lesion and/or maintenance of tumor marker level above the normal limits.
Time Frame: Maximum up to 18 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Percentage of participants | 56.9 | 66.7 | 50 | 100 | 62.7 | 55

41. Secondary Outcome: Disease Control Rate (DCR) at Month 12 and 18
Description: DCR at 12 and 18 months was defined as the percentage of participants with CR, PR or SD at 12 and at 18 months. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Persistence of one or more non-target lesion and/or maintenance of tumor marker level above the normal limits. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study or unequivocal progression of existing non-target lesions), taking as reference the smallest sum diameters while on study.
Time Frame: Month 12, 18
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Percentage of participants
  Month 12 | 76.5 | 80 | 50 | 100 | 78.4 | 75
  Month 18 | 76.5 | 80 | 50 | 100 | 78.4 | 75

42. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) Lung Cancer (LC) Module 13 Symptom Scales Scores at Baseline, Month 3, 6, 9, 12, 15 and 18
Description: EORTC QLQ-LC13 consisted of following symptom scales/items: coughing, haemoptysis, dyspnoea, dyspnoea when resting, dyspnoea when walking, dyspnoea when stairs, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts and pain relief after medication. The dyspnoea scale was only calculated if all three items had been answered. Some respondents ignore question "dyspnoea when stairs" because they never climbed stairs. Hence if item "dyspnoea when stairs" was missing then items "dyspnoea when resting" and "dyspnoea when walking" was used as single-item measures under item "dyspnoea". Transformed scores for each item ranged from 0 to 100, higher score is indicative of a higher response level (a high score for a symptom scale/item represents a high level of symptomatology/problems).
Time Frame: Baseline, Month 3, 6, 9, 12, 15, 18
Population: FFAS included all eligible participants (with known ALK or ROS1 gene rearrangement) who received at least 1 dose of Crizotinib. Here, "number analyzed" signifies participants evaluable for the specified rows.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Units on a scale
  Coughing: Baseline: number analyzed (Participants) | 46 | 11 | 2 | 2 | 45 | 16
  Coughing: Baseline | 33.30 [33.30 to 66.70] | 33.30 [0.00 to 33.30] | 16.65 [0.00 to 33.30] | 50.00 [0.00 to 100.00] | 33.30 [0.00 to 66.70] | 33.30 [0.00 to 33.30]
  Haemoptysis: Baseline: number analyzed (Participants) | 46 | 11 | 2 | 2 | 45 | 16
  Haemoptysis: Baseline | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Dyspnoea: Baseline: number analyzed (Participants) | 40 | 11 | 2 | 2 | 40 | 15
  Dyspnoea: Baseline | 22.20 [0.00 to 44.40] | 22.20 [11.10 to 55.60] | 11.10 [0.00 to 22.20] | 22.20 [22.20 to 22.20] | 22.20 [0.00 to 38.85] | 33.30 [11.10 to 44.40]
  Dyspnoea when resting: Baseline: number analyzed (Participants) | 45 | 11 | 2 | 2 | 44 | 16
  Dyspnoea when resting: Baseline | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 16.65]
  Dyspnoea when walking: Baseline: number analyzed (Participants) | 44 | 11 | 2 | 2 | 44 | 15
  Dyspnoea when walking: Baseline | 33.30 [0.00 to 66.70] | 33.30 [0.00 to 66.70] | 16.65 [0.00 to 33.30] | 33.30 [0.00 to 33.30] | 33.30 [0.00 to 50.00] | 33.30 [33.30 to 66.70]
  Dyspnoea when stairs: Baseline: number analyzed (Participants) | 41 | 11 | 2 | 2 | 41 | 15
  Dyspnoea when stairs: Baseline | 33.30 [0.00 to 66.70] | 33.30 [33.30 to 33.30] | 16.65 [0.00 to 33.30] | 33.30 [33.30 to 33.30] | 33.30 [0.00 to 66.70] | 33.30 [33.30 to 66.70]
  Sore mouth: Baseline: number analyzed (Participants) | 46 | 11 | 2 | 2 | 45 | 16
  Sore mouth: Baseline | 0 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Dysphagia: Baseline: number analyzed (Participants) | 46 | 11 | 1 | 2 | 44 | 16
  Dysphagia: Baseline | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00]
  Peripheral neuropathy: Baseline: number analyzed (Participants) | 46 | 11 | 2 | 2 | 45 | 16
  Peripheral neuropathy: Baseline | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 33.30] | 33.35 [0.00 to 66.70] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 16.65]
  Alopecia: Baseline: number analyzed (Participants) | 46 | 11 | 2 | 2 | 45 | 16
  Alopecia: Baseline | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Pain Chest: Baseline: number analyzed (Participants) | 46 | 11 | 2 | 2 | 45 | 16
  Pain Chest: Baseline | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 16.65 [0.00 to 33.30] | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 16.65]
  Pain Arm/Shoulders: Baseline: number analyzed (Participants) | 46 | 11 | 2 | 2 | 45 | 16
  Pain Arm/Shoulders: Baseline | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 33.30] | 16.65 [0.00 to 33.30] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00]
  Pain Other Parts: Baseline: number analyzed (Participants) | 43 | 11 | 2 | 2 | 43 | 15
  Pain Other Parts: Baseline | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] | 50.00 [33.30 to 66.70] | 0.00 [0.00 to 33.30] | 33.30 [0.00 to 33.30]
  Pain relief after medication: Baseline: number analyzed (Participants) | 16 | 4 | 1 | 1 | 14 | 8
  Pain relief after medication: Baseline | 66.70 [33.30 to 100.00] | 50.00 [33.30 to 83.35] | 33.30 [33.30 to 33.30] | 100.00 [100.00 to 100.00] | 66.70 [33.30 to 100.00] | 33.30 [33.30 to 83.35]
  Coughing: Month 3: number analyzed (Participants) | 34 | 12 | 1 | 2 | 36 | 13
  Coughing: Month 3 | 0.00 [0.00 to 33.30] | 16.65 [0.00 to 33.30] | 66.70 [66.70 to 66.70] | 16.65 [0.00 to 33.30] | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 33.30]
  Haemoptysis: Month 3: number analyzed (Participants) | 34 | 12 | 1 | 2 | 36 | 13
  Haemoptysis: Month 3 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 66.70 [66.70 to 66.70] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Dyspnoea: Month 3: number analyzed (Participants) | 33 | 11 | 1 | 2 | 34 | 13
  Dyspnoea: Month 3 | 11.10 [0.00 to 22.20] | 22.20 [11.10 to 44.40] | 66.70 [66.70 to 66.70] | 16.65 [0.00 to 33.30] | 11.10 [0.00 to 22.20] | 22.20 [11.10 to 33.30]
  Dyspnoea when resting: Month 3: number analyzed (Participants) | 34 | 12 | 1 | 2 | 36 | 13
  Dyspnoea when resting: Month 3 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 16.65] | 66.70 [66.70 to 66.70] | 16.65 [0.00 to 33.30] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Dyspnoea when walking: Month 3: number analyzed (Participants) | 34 | 12 | 1 | 2 | 36 | 13
  Dyspnoea when walking: Month 3 | 0.00 [0.00 to 33.30] | 33.30 [0.00 to 50.00] | 66.70 [66.70 to 66.70] | 16.65 [0.00 to 33.30] | 0.00 [0.00 to 33.30] | 33.30 [0.00 to 33.30]
  Dyspnoea when stairs: Month 3: number analyzed (Participants) | 33 | 11 | 1 | 2 | 34 | 13
  Dyspnoea when stairs: Month 3 | 33.30 [0.00 to 33.30] | 33.30 [33.30 to 66.70] | 66.70 [66.70 to 66.70] | 16.65 [0.00 to 33.30] | 33.30 [0.00 to 33.30] | 33.30 [0.00 to 33.30]
  Sore mouth: Month 3: number analyzed (Participants) | 33 | 12 | 1 | 2 | 36 | 12
  Sore mouth: Month 3 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Dysphagia: Month 3: number analyzed (Participants) | 33 | 12 | 1 | 2 | 36 | 12
  Dysphagia: Month 3 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 66.70 [66.70 to 66.70] | 16.65 [0.00 to 33.30] | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00]
  Peripheral neuropathy: Month 3: number analyzed (Participants) | 34 | 12 | 1 | 2 | 36 | 13
  Peripheral neuropathy: Month 3 | 0.00 [0.00 to 33.30] | 33.30 [0.00 to 33.30] | 66.70 [66.70 to 66.70] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 33.30]
  Alopecia: Month 3: number analyzed (Participants) | 32 | 12 | 1 | 2 | 35 | 12
  Alopecia: Month 3 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Pain chest: Month 3: number analyzed (Participants) | 34 | 12 | 1 | 2 | 36 | 13
  Pain chest: Month 3 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 66.70 [66.70 to 66.70] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 16.65] | 0.00 [0.00 to 0.00]
  Pain arm/shoulders: Month 3: number analyzed (Participants) | 34 | 12 | 1 | 2 | 36 | 13
  Pain arm/shoulders: Month 3 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 33.30 [33.30 to 33.30] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Pain other parts: Month 3: number analyzed (Participants) | 33 | 12 | 0 | 2 | 35 | 12
  Pain other parts: Month 3 | 0.00 [0.00 to 33.30] | 33.30 [0.00 to 33.30] |  | 16.65 [0.00 to 33.30] | 0.00 [0.00 to 33.30] | 33.30 [0.00 to 50.00]
  Pain relief after medication: Month 3: number analyzed (Participants) | 11 | 3 | 1 | 0 | 10 | 5
  Pain relief after medication: Month 3 | 33.30 [33.30 to 100.00] | 33.30 [33.30 to 33.30] | 66.70 [66.70 to 66.70] |  | 33.30 [33.30 to 33.30] | 66.70 [66.70 to 100.00]
  Coughing: Month 6: number analyzed (Participants) | 24 | 8 | 0 | 0 | 26 | 6
  Coughing: Month 6 | 0.00 [0.00 to 33.30] | 33.30 [0.00 to 33.30] |  |  | 33.30 [0.00 to 33.30] | 0.00 [0.00 to 33.30]
  Haemoptysis: Month 6:: number analyzed (Participants) | 24 | 8 | 0 | 0 | 26 | 6
  Haemoptysis: Month 6: | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Dyspnoea: Month 6: number analyzed (Participants) | 23 | 6 | 0 | 0 | 24 | 5
  Dyspnoea: Month 6 | 22.20 [0.00 to 33.30] | 22.20 [22.20 to 66.70] |  |  | 22.20 [0.00 to 33.30] | 33.30 [11.10 to 66.70]
  Dyspnoea when resting: Month 6: number analyzed (Participants) | 23 | 7 | 0 | 0 | 25 | 5
  Dyspnoea when resting: Month 6 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 66.70] |  |  | 0.00 [0.00 to 0.00] | 33.30 [0.00 to 33.30]
  Dyspnoea when walking: Month 6: number analyzed (Participants) | 24 | 7 | 0 | 0 | 25 | 6
  Dyspnoea when walking: Month 6 | 16.65 [0.00 to 33.30] | 33.30 [33.30 to 66.70] |  |  | 33.30 [0.00 to 33.30] | 16.65 [0.00 to 66.70]
  Dyspnoea when stairs: Month 6: number analyzed (Participants) | 24 | 8 | 0 | 0 | 26 | 6
  Dyspnoea when stairs: Month 6 | 33.30 [0.00 to 50.00] | 33.30 [33.30 to 66.65] |  |  | 33.30 [0.00 to 33.30] | 33.30 [33.30 to 66.70]
  Sore mouth: Month 6: number analyzed (Participants) | 24 | 7 | 0 | 0 | 25 | 6
  Sore mouth: Month 6 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Dysphagia: Month 6: number analyzed (Participants) | 23 | 8 | 0 | 0 | 26 | 5
  Dysphagia: Month 6 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.30] |  |  | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00]
  Peripheral neuropathy: Month 6: number analyzed (Participants) | 24 | 6 | 0 | 0 | 24 | 6
  Peripheral neuropathy: Month 6 | 33.30 [0.00 to 50.00] | 33.30 [0.00 to 33.30] |  |  | 33.30 [0.00 to 33.30] | 16.65 [0.00 to 66.70]
  Alopecia: Month 6: number analyzed (Participants) | 24 | 7 | 0 | 0 | 25 | 6
  Alopecia: Month 6 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.30] |  |  | 0.00 [0.00 to 0.00] | 16.65 [0.00 to 33.30]
  Pain chest: Month 6: number analyzed (Participants) | 24 | 7 | 0 | 0 | 25 | 6
  Pain chest: Month 6 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Pain arm/shoulders: Month 6: number analyzed (Participants) | 24 | 8 | 0 | 0 | 26 | 6
  Pain arm/shoulders: Month 6 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Pain other parts: Month 6: number analyzed (Participants) | 24 | 7 | 0 | 0 | 25 | 6
  Pain other parts: Month 6 | 0.00 [0.00 to 66.70] | 0.00 [0.00 to 66.70] |  |  | 0.00 [0.00 to 66.70] | 0.00 [0.00 to 66.70]
  Pain relief after medication: Month 6: number analyzed (Participants) | 7 | 2 | 0 | 0 | 8 | 1
  Pain relief after medication: Month 6 | 33.30 [0.00 to 33.30] | 50.00 [0.00 to 100.00] |  |  | 33.30 [0.00 to 33.30] | 100.00 [100.00 to 100.00]
  Coughing: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Coughing: Month 9 | 0.00 [0.00 to 33.30] | 33.30 [0.00 to 33.30] |  |  | 33.30 [0.00 to 33.30] | 16.65 [0.00 to 33.30]
  Haemoptysis: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Haemoptysis: Month 9 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Dyspnoea: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Dyspnoea: Month 9 | 22.20 [0.00 to 33.30] | 38.85 [22.20 to 55.60] |  |  | 22.20 [0.00 to 44.40] | 27.75 [16.65 to 44.45]
  Dyspnoea when resting: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Dyspnoea when resting: Month 9 | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 16.65]
  Dyspnoea when walking: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Dyspnoea when walking: Month 9 | 33.30 [0.00 to 33.30] | 50.00 [33.30 to 66.70] |  |  | 33.30 [0.00 to 66.70] | 33.30 [16.65 to 50.00]
  Dyspnoea when stairs: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Dyspnoea when stairs: Month 9 | 33.30 [0.00 to 33.30] | 66.70 [33.30 to 66.70] |  |  | 33.30 [0.00 to 66.70] | 33.30 [33.30 to 66.65]
  Sore mouth: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Sore mouth: Month 9 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Dysphagia: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Dysphagia: Month 9 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Peripheral neuropathy: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Peripheral neuropathy: Month 9 | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 33.30] |  |  | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 16.65]
  Alopecia: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Alopecia: Month 9 | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 16.65]
  Pain chest: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Pain chest: Month 9 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Pain arm/shoulders: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Pain arm/shoulders: Month 9 | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 16.65]
  Pain other parts: Month 9: number analyzed (Participants) | 19 | 6 | 0 | 0 | 21 | 4
  Pain other parts: Month 9 | 0.00 [0.00 to 66.70] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 66.70] | 0.00 [0.00 to 50.00]
  Pain relief after medication: Month 9: number analyzed (Participants) | 6 | 3 | 0 | 0 | 8 | 1
  Pain relief after medication: Month 9 | 33.30 [0.00 to 100.00] | 33.30 [33.30 to 100.00] |  |  | 33.30 [16.65 to 66.65] | 100.00 [100.00 to 100.00]
  Coughing: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Coughing: Month 12 | 0.00 [0.00 to 33.30] | 16.65 [0.00 to 33.30] |  |  | 16.65 [0.00 to 33.30] | 0.00 [0.00 to 16.65]
  Haemoptysis: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Haemoptysis: Month 12 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Dyspnoea: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Dyspnoea: Month 12 | 33.30 [5.55 to 33.30] | 33.30 [27.75 to 50.00] |  |  | 27.75 [5.55 to 44.45] | 33.30 [33.30 to 33.30]
  Dyspnoea when resting: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Dyspnoea when resting: Month 12 | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 16.65] |  |  | 0.00 [0.00 to 16.65] | 16.65 [0.00 to 33.30]
  Dyspnoea when walking: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Dyspnoea when walking: Month 12 | 33.30 [0.00 to 66.70] | 33.30 [33.30 to 66.65] |  |  | 33.30 [0.00 to 66.70] | 33.30 [33.30 to 50.00]
  Dyspnoea when stairs: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Dyspnoea when stairs: Month 12 | 33.30 [0.00 to 33.30] | 50.00 [33.30 to 83.35] |  |  | 33.30 [0.00 to 66.65] | 33.30 [33.30 to 50.00]
  Sore mouth: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Sore mouth: Month 12 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Dysphagia: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Dysphagia: Month 12 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Peripheral neuropathy: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Peripheral neuropathy: Month 12 | 0.0 [0.0 to 33.30] | 0.0 [0.0 to 16.65] |  |  | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00]
  Alopecia: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Alopecia: Month 12 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Pain Chest: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Pain Chest: Month 12 | 0.00 [0.00 to 16.65] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 16.65] | 0.00 [0.00 to 0.00]
  Pain Arm/Shoulders: Month 12: number analyzed (Participants) | 16 | 4 | 0 | 0 | 16 | 4
  Pain Arm/Shoulders: Month 12 | 0.00 [0.00 to 16.65] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 16.65] | 0.00 [0.00 to 0.00]
  Pain Other Parts: Month 12: number analyzed (Participants) | 15 | 4 | 0 | 0 | 15 | 4
  Pain Other Parts: Month 12 | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 50.00]
  Pain relief after medication: Month 12: number analyzed (Participants) | 3 | 3 | 0 | 0 | 5 | 1
  Pain relief after medication: Month 12 | 33.30 [0.00 to 100.00] | 100.00 [33.30 to 100.00] |  |  | 33.30 [33.30 to 100.00] | 100.00 [100.00 to 100.00]
  Coughing: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Coughing: Month 15 | 16.65 [0.00 to 33.30] | 33.30 [33.30 to 100.00] |  |  | 33.30 [0.00 to 33.30] | 50.00 [0.00 to 100.00]
  Haemoptysis: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Haemoptysis: Month 15 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Dyspnoea: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Dyspnoea: Month 15 | 16.65 [0.00 to 27.75] | 66.70 [22.20 to 66.70] |  |  | 22.20 [0.00 to 33.30] | 33.35 [0.00 to 66.70]
  Dyspnoea when resting: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Dyspnoea when resting: Month 15 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.30] |  |  | 0.00 [0.00 to 0.00] | 16.65 [0.00 to 33.30]
  Dyspnoea when walking: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Dyspnoea when walking: Month 15 | 16.65 [0.00 to 33.30] | 66.70 [33.30 to 100.00] |  |  | 33.30 [0.00 to 33.30] | 33.35 [0.00 to 66.70]
  Dyspnoea when stairs: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Dyspnoea when stairs: Month 15 | 16.65 [0.00 to 33.30] | 100.00 [33.30 to 100.00] |  |  | 33.30 [0.00 to 33.30] | 50.00 [0.00 to 100.00]
  Sore mouth: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Sore mouth: Month 15 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.30] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Dysphagia: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Dysphagia: Month 15 | 0.00 [0.00 to 0.00] | 33.30 [0.00 to 66.70] |  |  | 0.00 [0.00 to 0.00] | 16.65 [0.00 to 33.30]
  Peripheral neuropathy: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Peripheral neuropathy: Month 15 | 16.65 [0.00 to 50.00] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00]
  Alopecia: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Alopecia: Month 15 | 0.00 [0.00 to 16.65] | 0.00 [0.00 to 33.30] |  |  | 0.00 [0.00 to 0.00] | 16.65 [0.00 to 33.30]
  Pain Chest: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Pain Chest: Month 15 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Pain Arm/Shoulders: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Pain Arm/Shoulders: Month 15 | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00]
  Pain Other Parts: Month 15: number analyzed (Participants) | 12 | 3 | 0 | 0 | 13 | 2
  Pain Other Parts: Month 15 | 0.00 [0.00 to 16.65] | 66.70 [33.30 to 66.70] |  |  | 0.00 [0.00 to 33.30] | 33.35 [0.00 to 66.70]
  Pain relief after medication: Month 15: number analyzed (Participants) | 0 | 3 | 0 | 0 | 2 | 1
  Pain relief after medication: Month 15 |  | 33.30 [33.30 to 100.00] |  |  | 66.65 [33.30 to 100.00] | 33.30 [33.30 to 33.30]
  Coughing: Month 18: number analyzed (Participants) | 8 | 2 | 0 | 0 | 9 | 1
  Coughing: Month 18 | 33.30 [0.00 to 50.00] | 50.00 [33.30 to 66.70] |  |  | 33.30 [0.00 to 33.30] | 100.00 [100.00 to 100.00]
  Haemoptysis: Month 18: number analyzed (Participants) | 8 | 2 | 0 | 0 | 9 | 1
  Haemoptysis: Month 18 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Dyspnoea: Month 18: number analyzed (Participants) | 7 | 1 | 0 | 0 | 7 | 1
  Dyspnoea: Month 18 | 33.30 [22.20 to 66.70] | 55.60 [55.60 to 55.60] |  |  | 33.30 [22.20 to 55.60] | 66.70 [66.70 to 66.70]
  Dyspnoea when resting: Month 18: number analyzed (Participants) | 8 | 2 | 0 | 0 | 9 | 1
  Dyspnoea when resting: Month 18 | 16.65 [0.00 to 33.30] | 33.35 [0.00 to 66.70] |  |  | 0.00 [0.00 to 33.30] | 33.30 [33.30 to 33.30]
  Dyspnoea when walking: Month 18: number analyzed (Participants) | 8 | 1 | 0 | 0 | 8 | 1
  Dyspnoea when walking: Month 18 | 33.30 [16.65 to 66.70] | 66.70 [66.70 to 66.70] |  |  | 33.30 [16.65 to 66.70] | 66.70 [66.70 to 66.70]
  Dyspnoea when stairs: Month 18: number analyzed (Participants) | 7 | 2 | 0 | 0 | 8 | 1
  Dyspnoea when stairs: Month 18 | 33.30 [33.30 to 100.00] | 66.65 [33.30 to 100.00] |  |  | 33.30 [33.30 to 83.35] | 100.00 [100.00 to 100.00]
  Sore mouth: Month 18: number analyzed (Participants) | 8 | 2 | 0 | 0 | 9 | 1
  Sore mouth: Month 18 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Dysphagia: Month 18: number analyzed (Participants) | 8 | 2 | 0 | 0 | 9 | 1
  Dysphagia: Month 18 | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 33.30 [33.30 to 33.30]
  Peripheral neuropathy: Month 18: number analyzed (Participants) | 8 | 2 | 0 | 0 | 9 | 1
  Peripheral neuropathy: Month 18 | 33.30 [0.00 to 50.00] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 33.30] | 33.30 [33.30 to 33.30]
  Alopecia: Month 18: number analyzed (Participants) | 8 | 2 | 0 | 0 | 9 | 1
  Alopecia: Month 18 | 33.30 [0.00 to 33.30] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 33.30] | 66.70 [66.70 to 66.70]
  Pain Chest: Month 18: number analyzed (Participants) | 8 | 2 | 0 | 0 | 9 | 1
  Pain Chest: Month 18 | 16.65 [0.00 to 33.30] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 33.30] | 33.30 [33.30 to 33.30]
  Pain Arm/Shoulders: Month 18: number analyzed (Participants) | 8 | 2 | 0 | 0 | 9 | 1
  Pain Arm/Shoulders: Month 18 | 0.00 [0.00 to 16.65] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 0.00] | 33.30 [33.30 to 33.30]
  Pain Other Parts: Month 18: number analyzed (Participants) | 7 | 2 | 0 | 0 | 8 | 1
  Pain Other Parts: Month 18 | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00] |  |  | 0.00 [0.00 to 33.30] | 0.00 [0.00 to 0.00]
  Pain relief after medication: Month 18: number analyzed (Participants) | 4 | 1 | 0 | 0 | 5 | 0
  Pain relief after medication: Month 18 | 50.00 [33.30 to 83.35] | 33.30 [33.30 to 33.30] |  |  | 33.30 [33.30 to 66.70] |

43. Secondary Outcome: Time to Median Progression Free Survival (Months) With Its 95%CI
Description: PFS was defined as the time between the treatment start (date of the first Crizotinib intake) and the date of the first disease progression or the all-cause death. Participants who did not progress or were still alive at the end of the study or at the date of cut-off were censored at the last disease evaluation date.
Time Frame: 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Months | 9.2 [6.2 to 13.7] | 9.2 [5.8 to NA] — Unable to estimate the 95% upper limit due to insufficient number of participants with events. | NA [NA to NA] — Unable to estimate due to insufficient number of participants with events. | NA [NA to NA] — Unable to estimate due to insufficient number of participants with events. | 9.4 [7.0 to 16.4] | 6.6 [4.3 to 14.3]

44. Secondary Outcome: 18-Month Overall Survival (OS) Rate (95%CI)
Description: OS was defined as the time from the date of first dose of study drug to the date of death due to any cause. Participants last known to be alive were censored at the date of last contact. 18-month OS rates was assessed by Kaplan-Meier method with right censoring.
Time Frame: 18 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20
Percentage of participants | 61.5 [46.3 to 73.5] | 77.8 [45.5 to 92.3] | NA [NA to NA] — Unable to estimate due to insufficient number of participants with events. | NA [NA to NA] — Unable to estimate due to insufficient number of participants with events. | 77.5 [63.0 to 86.9] | 40.5 [18.1 to 62.0]

45. Secondary Outcome: Number of Participants Per Morisky Score Classification at Month 3, 6, 9, 12, 15 and 18
Description: Compliance to study drug was evaluated using Morisky score. The questionnaire consisted of 4 questions in which the scale was 0 for "yes" (indicating poor compliance) and 1 for "no" (indicating good compliance). The items were summed to give a range of scores from 0 to 4. A score of 4 indicated high compliance, 2-3 indicated medium compliance and 0-1 indicated low compliance.
Time Frame: Month 3, 6, 9, 12, 15 and 18
Population: Safety population included all enrolled participants who received at least 1 dose of Crizotinib. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Groups:
- Crizotinib: ALK+ NSCLC: Participants aged >=18 years, followed up for locally advanced (stage IIIB not suitable for radiotherapy) or metastatic (stage IV) ALK+ NSCLC initiating (or having initiated in previous 3 months) treatment with crizotinib regardless of the line of treatment were sequentially included in this observational, descriptive, longitudinal, multicentre, retroprospective study. The participants received crizotinib as per normal routine healthcare practice in real world. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
- Crizotinib: ROS+ NSCLC: Participants aged >=18 years, followed up for locally advanced (stage IIIB not suitable for radiotherapy) or metastatic (stage IV) ALK+ NSCLC initiating (or having initiated in previous 3 months) treatment with crizotinib regardless of line of treatment were sequentially included in this observational, descriptive, longitudinal, multicentre, retroprospective study. The participants received crizotinib as per normal routine healthcare practice in real world. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC | Participants With Unknown Gene Rearrangement
Number analyzed (Participants) | 48 | 14 | 2 | 3 | 48 | 19 | 0
Participants
  Month 3: Missing | 13 | 2 | 1 | 1 | 11 | 6 |
  Month 3: Morisky score 1 | 1 | 0 | 0 | 0 | 0 | 1 |
  Month 3: Morisky score 2 | 2 | 0 | 0 | 0 | 1 | 1 |
  Month 3: Morisky score 3 | 4 | 2 | 0 | 0 | 6 | 0 |
  Month 3: Morisky score 4 | 28 | 10 | 1 | 2 | 30 | 11 |
  Month 6: number analyzed (Participants) | 38 | 12 | 1 | 3 | 40 | 14 | 0
  Month 6: Missing | 14 | 4 | 1 | 3 | 14 | 8 |
  Month 6: Morisky score 1 | 0 | 0 | 0 | 0 | 0 | 0 |
  Month 6: Morisky score 2 | 0 | 1 | 0 | 0 | 1 | 0 |
  Month 6: Morisky score 3 | 5 | 1 | 0 | 0 | 5 | 1 |
  Month 6: Morisky score 4 | 19 | 6 | 0 | 0 | 20 | 5 |
  Month 9: number analyzed (Participants) | 29 | 7 | 1 | 1 | 28 | 10 | 0
  Month 9: Missing | 10 | 1 | 1 | 1 | 7 | 6 |
  Month 9: Morisky score 1 | 0 | 0 | 0 | 0 | 0 | 0 |
  Month 9: Morisky score 2 | 0 | 0 | 0 | 0 | 0 | 0 |
  Month 9: Morisky score 3 | 2 | 2 | 0 | 0 | 3 | 1 |
  Month 9: Morisky score 4 | 17 | 4 | 0 | 0 | 18 | 3 |
  Month 12: number analyzed (Participants) | 24 | 7 | 1 | 1 | 26 | 7 | 0
  Month 12: Missing | 8 | 3 | 1 | 1 | 10 | 3 |
  Month 12: Morisky score 1 | 0 | 0 | 0 | 0 | 0 | 0 |
  Month 12: Morisky score 2 | 0 | 0 | 0 | 0 | 0 | 0 |
  Month 12: Morisky score 3 | 4 | 1 | 0 | 0 | 4 | 1 |
  Month 12: Morisky score 4 | 12 | 3 | 0 | 0 | 12 | 3 |
  Month 15: number analyzed (Participants) | 17 | 7 | 1 | 0 | 22 | 3 | 0
  Month 15: Missing | 5 | 4 | 1 |  | 9 | 1 |
  Month 15: Morisky score 1 | 0 | 0 | 0 |  | 0 | 0 |
  Month 15: Morisky score 2 | 0 | 0 | 0 |  | 0 | 0 |
  Month 15: Morisky score 3 | 2 | 0 | 0 |  | 2 | 0 |
  Month 15: Morisky score 4 | 10 | 3 | 0 |  | 11 | 2 |
  Month 18: number analyzed (Participants) | 16 | 5 | 1 | 0 | 18 | 4 | 0
  Month 18: Missing | 8 | 3 | 1 |  | 9 | 3 |
  Month 18: Morisky score 1 | 0 | 0 | 0 |  | 0 | 0 |
  Month 18: Morisky score 2 | 0 | 0 | 0 |  | 0 | 0 |
  Month 18: Morisky score 3 | 1 | 0 | 0 |  | 1 | 0 |
  Month 18: Morisky score 4 | 7 | 2 | 0 |  | 8 | 1 |

46. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Serious AE: any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and all Non-SAEs.
Time Frame: Up to maximum of 18 months
Population: Safety population included all enrolled participants who received at least 1 dose of Crizotinib.
Measure: Count of Participants; unit: Participants
Groups:
- Crizotinib: Other Line of Treatment: Participants included in this arm were treated with crizotinib as other line of treatment for advanced or metastatic NSCLC with ALK or ROS gene rearrangement, per normal routine medical care in real world practices. The participants were followed until the participant's death or early withdrawal from the study for another reason (up to maximum of 18 months).
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Crizotinib: ALK+ NSCLC | Crizotinib: ROS+ NSCLC | Participants With Unknown Gene Rearrangement
Number analyzed (Participants) | 51 | 15 | 2 | 3 | 51 | 20 | 2
Participants
  AE | 49 | 13 | 2 | 3 | 47 | 20 | 0
  SAE | 32 | 6 | 0 | 1 | 25 | 14 | 0

ADVERSE EVENTS:
Time Frame: Up to maximum of 18 months
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis set included all enrolled participants who received at least 1 dose of Crizotinib.
Arm/Group | Crizotinib: First Line of Treatment | Crizotinib: Second Line of Treatment | Crizotinib: Third Line of Treatment | Crizotinib: Other Line of Treatment | Participants With ALK Gene Rearrangement | Participants With ROS1 Gene Rearrangement | Participants With Unknown Gene Rearrangement
All-Cause Mortality (participants affected / at risk) | 21/51 | 3/15 | 0/2 | 0/3 | 13/51 | 11/20 | 0/2
Serious Adverse Events (participants affected / at risk) | 32/51 | 6/15 | 0/2 | 1/3 | 25/51 | 14/20 | 0/2
Other Adverse Events (participants affected / at risk) | 42/51 | 12/15 | 2/2 | 3/3 | 43/51 | 16/20 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib: First Line of Treatment (N=51) | Crizotinib: Second Line of Treatment (N=15) | Crizotinib: Third Line of Treatment (N=2) | Crizotinib: Other Line of Treatment (N=3) | Participants With ALK Gene Rearrangement (N=51) | Participants With ROS1 Gene Rearrangement (N=20) | Participants With Unknown Gene Rearrangement (N=2)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 9 | 0 | 0 | 0 | 3 | 6 | 0
DEATH (General disorders) | 3 | 2 | 0 | 0 | 4 | 1 | 0
ASTHENIA (General disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
CHEST PAIN (General disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
CONDITION AGGRAVATED (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 2 | 1 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1 | 2 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 2 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
INTESTINAL INFARCTION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 0 | 0 | 0 | 3 | 6 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0 | 0
CANDIDA INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
LYMPHANGITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
PNEUMOCYSTIS JIROVECII (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
UROSEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
TACHYARRHYTHMIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
CEREBRAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
CEREBRAL VENOUS THROMBOSIS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
NEURALGIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 3 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
PRODUCT DISPENSING ERROR (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
HEPATOTOXICITY (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
DISABILITY (Social circumstances) | 1 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib: First Line of Treatment (N=51) | Crizotinib: Second Line of Treatment (N=15) | Crizotinib: Third Line of Treatment (N=2) | Crizotinib: Other Line of Treatment (N=3) | Participants With ALK Gene Rearrangement (N=51) | Participants With ROS1 Gene Rearrangement (N=20) | Participants With Unknown Gene Rearrangement (N=2)
NAUSEA (Gastrointestinal disorders) | 18 | 4 | 1 | 2 | 18 | 7 | 0
DIARRHOEA (Gastrointestinal disorders) | 20 | 2 | 1 | 2 | 19 | 6 | 0
VOMITING (Gastrointestinal disorders) | 11 | 2 | 1 | 1 | 11 | 4 | 0
CONSTIPATION (Gastrointestinal disorders) | 9 | 1 | 0 | 0 | 6 | 4 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 2 | 0 | 1 | 6 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 4 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 2 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
APHTHOUS ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
FUNCTIONAL GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
GASTRIC DISORDER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 14 | 2 | 0 | 1 | 10 | 7 | 0
ASTHENIA (General disorders) | 6 | 4 | 1 | 0 | 8 | 3 | 0
FATIGUE (General disorders) | 5 | 1 | 1 | 0 | 6 | 1 | 0
CHEST PAIN (General disorders) | 2 | 0 | 1 | 0 | 2 | 1 | 0
CREPITATIONS (General disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0
FACE OEDEMA (General disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0
PYREXIA (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
ADVERSE EVENT (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
CONDITION AGGRAVATED (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
DISCOMFORT (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
MASS (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
MUCOSAL DRYNESS (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
PAIN (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 7 | 0 | 1 | 0 | 7 | 1 | 0
DYSGEUSIA (Nervous system disorders) | 5 | 1 | 0 | 0 | 6 | 0 | 0
TASTE DISORDER (Nervous system disorders) | 2 | 0 | 0 | 1 | 2 | 1 | 0
HEADACHE (Nervous system disorders) | 2 | 1 | 0 | 0 | 3 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0
DYSAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
TREMOR (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
HEAD DISCOMFORT (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
HYPERAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
HYPERSOMNIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
MOTOR DYSFUNCTION (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
TENSION HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
VISUAL IMPAIRMENT (Eye disorders) | 15 | 3 | 1 | 0 | 15 | 4 | 0
VISION BLURRED (Eye disorders) | 2 | 1 | 0 | 0 | 3 | 0 | 0
PHOTOPSIA (Eye disorders) | 2 | 1 | 0 | 0 | 3 | 0 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 3 | 0 | 0 | 0 | 3 | 0 | 0
CHALAZION (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
CATARACT (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
CHROMATOPSIA (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
VITREOUS FLOATERS (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
WEIGHT DECREASED (Investigations) | 4 | 1 | 0 | 0 | 3 | 2 | 0
WEIGHT INCREASED (Investigations) | 4 | 0 | 0 | 0 | 2 | 2 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 0 | 0 | 1 | 3 | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0 | 0 | 1 | 2 | 1 | 0
TRANSAMINASES INCREASED (Investigations) | 2 | 0 | 0 | 1 | 3 | 0 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 | 0 | 0 | 0 | 1 | 1 | 0
BLOOD COUNT ABNORMAL (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
BREATH SOUNDS ABNORMAL (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
GAMMAGLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
LIPASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
VITAMIN D DECREASED (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 1 | 0 | 6 | 4 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0 | 1 | 4 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 3 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 | 4 | 0 | 1 | 10 | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0
FOOD AVERSION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 2 | 0 | 1 | 4 | 2 | 0
ANAEMIA (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 2 | 1 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 4 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 2 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
BONE LESION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
ORAL HERPES (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
TINEA VERSICOLOUR (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
SUPERINFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 4 | 0 | 0 | 0 | 1 | 3 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
PRURIGO (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 4 | 0 | 0 | 0 | 4 | 0 | 0
MENIERE'S DISEASE (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
TINNITUS (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
CARDIAC DISORDER (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
HOT FLUSH (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
LYMPHOEDEMA (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
HEPATIC CYTOLYSIS (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 2 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
HEPATOTOXICITY (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0
MIXED ANXIETY AND DEPRESSIVE DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
SLEEP DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT03718117/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03718117/SAP_001.pdf